CLINICAL TRIAL: NCT00294268
Title: A Maintenance-Oriented Cognitive Behavioural Therapy in the Treatment of Obesity
Brief Title: Cognitive Behavioural Therapy for Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Dr Elizabeth Rieger, University of Sydney
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: erie8202
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-07

CONDITIONS: Obesity
Keywords: obesity; CBT; motivational enhancement therapy; weight loss maintenance
MeSH Terms: conditions — Obesity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): 20 weekly sessions of CBT integrated with motivational enhancement strategies
  Interventions: Behavioral: cognitive behavioural therapy

INTERVENTIONS:
Behavioral: cognitive behavioural therapy — 20 weekly sessions of CBT integrated with motivational enhancement strategies

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a cognitive behavioural treatment (CBT) designed to help obese patients lose weight and to maintain their weight losses over time. It is hypothesized that CBT will result in greater sustained weight loss.

DETAILED DESCRIPTION:
The primary aim of the present study is to improve the maintenance of weight loss, and hence the physical, psychological and social well-being, of obese patients who have sought weight loss treatment. To do so, it will implement a cognitive-behavioural treatment (CBT) with motivational enhancement strategies specifically designed to target weight maintenance. It is hypothesized that the maintenance-oriented CBT approach will result in sustained weight loss, as well as improved physical, psychological and social well-being.

ELIGIBILITY:
Inclusion Criteria:

* The participants will be recruited from among patients referred to the Metabolism and Obesity Service of Royal Prince Alfred Hospital.
* The inclusion criteria include: 18-65 years of age and a body mass index (BMI: kg/m2) between 30-45.

Exclusion Criteria:

* psychiatric conditions (i.e., current psychosis, severe depression, mental retardation, and drug or alcohol abuse)
* or physical conditions (i.e., significant hepatic or renal dysfunction and significant cardiovascular disease such as heart failure, stroke and transient ischaemic attacks) that would preclude full participation in the study;
* current treatment for obesity;
* current treatments known to affect eating or weight (e.g., medications);
* pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Weight | baseline, post-treatment, one-year follow-up

SECONDARY OUTCOMES:
obesity-specific quality of life, mood disturbance, eating disturbance, cognitive disturbance | baseline, post-treatment, one-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Rieger, PhD, Principal Investigator — University of Sydney
Locations (1):
- Metabolism and Obesity Services, Royal Prince Alfred Hospital, Sydney, New South Wales, Australia